CLINICAL TRIAL: NCT01739335
Title: Novel Therapeutics in PTSD: A Randomized Clinical Trial of Mifepristone
Brief Title: Novel Therapeutics in Posttraumatic Stress Disorder (PTSD): A Randomized Clinical Trial of Mifepristone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBA-04-11S; NCT01946685 (obsolete NCT alias)
Record Dates: First submitted 2012-11-15; First posted 2012-12-03 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Mifepristone; Veterans; Clinical Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mifepristone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mifepristone (Experimental): 'Mifepristone Oral Tablet [Korlym] (2 x 300mg =600 mg total, once daily, at bedtime) for 7 days
  Interventions: Drug: Mifepristone Oral Tablet [Korlym]
- Placebo (Placebo Comparator): Placebo Oral tablet (2 sugar pills, once daily, at bedtime) for 7 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mifepristone Oral Tablet [Korlym] — 2 Mifepristone 300 MG Oral Tablets once daily (600mg total) for 7 days
  Other Names: Korlym
  Arms: Mifepristone
Drug: Placebo Oral Tablet — 2 Placebo Oral Tablets once daily for 7 days
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Posttraumatic stress disorder (PTSD) is a common and disabling psychiatric disorder for Veterans. Left untreated or under-treated, it can become a chronic condition associated with significant distress, depression, aggression, family disruption, substance abuse and an increased risk of morbidity and mortality. Considerable advances were made in the treatment of PTSD in recent years; however, psychopharmacological treatments have been shown to be largely ineffective for Veterans with PTSD.

To address this gap, this proposal seeks to test an innovative treatment approach in PTSD - pharmacological manipulation of the body's major stress system (the hypothalamic-pituitary-adrenal (HPA) axis) with mifepristone. At high doses mifepristone is a glucocorticoid receptor (GR) antagonist with peripheral and central nervous system effects, making it a compound of interest in the treatment of stress related disorders. There is abundant evidence of enhanced GR sensitivity in Veterans with PTSD which is thought to underlie some of the symptoms of PTSD and associated disturbances in mood and cognition. There is also evidence that short-term mifepristone treatment has sustained beneficial effects on mood, cognition and sleep disturbance in some neuropsychiatric conditions (major depression, bipolar disorder, primary insomnia). The purpose of the study is to examine the effects of mifepristone to determine if it is efficacious in improving PTSD symptoms and associated clinical outcomes.

To achieve these objectives, the investigators propose to conduct a Phase IIa, multi-site, double-blind, placebo controlled trial of mifepristone in male Veteran outpatients with chronic PTSD through the VA's Cooperative Clinical Trial Award program. The investigators propose to enroll 90 subjects at multiple VA sites based on an estimated attrition rate of 20%. Eligible Veterans will be randomly assigned to the treatment of mifepristone (600 mg/day) or placebo for one week and followed for up to three months. The investigators will also describe the effects of mifepristone on several other clinical parameters including PTSD symptomology, depression severity, sleep quality, and functional impairment. Several measures of neuroendocrine functioning will also be obtained to explore the relationship of plasma cortisol and adrenocorticotropic hormone (ACTH) levels to clinical response and the time to addition of rescue medications.

DETAILED DESCRIPTION:
Novel approaches to the treatment of post traumatic stress disorder (PTSD) in Veterans are urgently needed. This proposal seeks to test an innovative approach, one that involves careful pharmacological manipulation of the body's major stress system, the hypothalamic-pituitary-adrenal (HPA) axis, using one dose of the FDA-approved drug, mifepristone (600 mg/day).

The rationale for a treatment trial of mifepristone in PTSD is based on the wealth of knowledge available about persistent alterations of the HPA axis in PTSD and their interactions with the central and autonomic nervous system and the immune system. The most consistent HPA axis findings in PTSD, taken together, suggest there is increased sensitivity to the effects of glucocorticoids in the presence of increased central activation of the HPA axis. Among the most replicated neuroendocrine findings have been of elevated levels of corticotropin-releasing factor (CRF) in the cerebrospinal fluid (CSF), an exaggerated cortisol response to emotional stressors, and an exaggerated suppression of cortisol to the synthetic glucocorticoid dexamethasone (DEX). The earliest studies of the effects of dexamethasone (DEX) using the standard 1.0 mg dose, found that PTSD, unlike major depression, was not associated with higher rates of cortisol non-suppression and there was a trend for lower cortisol levels post-DEX in PTSD. A lower dose (0.5 mg) was employed to test the hypothesis of enhanced suppression of cortisol to DEX in Vietnam Veterans with PTSD, which was confirmed. Since then, with few exceptions, greater suppression of cortisol to low-dose DEX has been found in PTSD subjects, compared to unexposed and/or trauma-exposed controls without PTSD, in diverse samples, including samples of persons exposed to combat, natural disasters, domestic violence, the Holocaust, and childhood physical and sexual abuse. Furthermore, the extent of cortisol suppression is associated with PTSD symptom severity. The finding of a greater down-regulation of lymphocyte GR post-DEX suggests that the dexamethasone suppression test (DST) findings may be attributable to more responsive glucocorticoid receptors. More recent studies have demonstrated increased suppression of ACTH to DEX confirming increased glucocorticoid responsivity at the level of the pituitary. The studies of the effects of DEX on HPA axis activity suggest there is enhanced negative feedback inhibition of the HPA axis in PTSD. Such inhibition could help to explain why despite evidence of central HPA axis activation and an exaggerated response of cortisol to stressors and to ACTH stimulation in PTSD, 24-hour basal cortisol levels are not typically elevated and indeed are even sometimes low.

Mifepristone is a selective type II glucocorticoid receptor antagonist with a favorable safety profile. It binds to the same site as the synthetic glucocorticoid dexamethasone and blocks the negative feedback control of cortisol on the pituitary. Thus, mifepristone, because it directly antagonizes the glucocorticoid receptor, which has been found to be more sensitive in PTSD in several models, is ideally suited for use in determining the pathophysiological significance of increased glucocorticoid receptor sensitivity in PTSD and whether its attenuation is of therapeutic value.

The investigators propose to study the clinical, neuropsychological, and neuroendocrine effects of short-term treatment with one dose of mifepristone (600 mg/day) in a well-characterized sample of Veterans with PTSD to determine if this treatment is effective in achieving a clinical response in PTSD, as well as improving clinical symptoms and quality of life. Furthermore, if pulse therapy with mifepristone has sustained effects, it holds out the promise of a very different approach to pharmacological treatment, one that may be preferable to Veterans who do not want to be on psychopharmacological treatments continuously or long-term.

Primary Objective

1. To determine whether 600 mg of mifepristone daily for one week in male Veterans with chronic PTSD yields a sufficiently high proportion of clinical responders after one month to warrant more extensive and definitive research.

Secondary Objectives

1. To study the trajectories of Clinician Administered PTSD Scale (CAPS)(CAPS) (past week symptom status) scores over the study duration for mifepristone and placebo.
2. To determine the effect of mifepristone compared to placebo on the time to addition of rescue medication.
3. To determine if a Phase III study is justified.
4. To compare adverse events (AEs) and serious adverse events (SAEs) in the two groups.

This Phase IIa clinical trial seeks to enroll 90 eligible male Veterans (assumes 20% attrition rate) with chronic PTSD. Participants will be randomly assigned to treatment with 600 mg/day mifepristone or placebo for one week and assessed for clinical outcomes at one and three months follow-up. Eligibility will be based on the inclusion and exclusion criteria which are enumerated below and in the Human Participants section. The investigators plan to include male Veterans with chronic PTSD who are not receiving psychotropic medication. The inclusion and exclusion criteria were selected in order to include as representative a sample as possible while also addressing safety concerns. Veterans who are actively suicidal as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) or who have attempted suicide within the past two years will be excluded. (If suicidality is identified, the necessary steps will be taken to ensure the appropriate clinical care is provided, and the local suicide prevention policies implemented.) Veterans with adrenal insufficiency will be excluded, as will Veterans with other major medical or neurological illnesses, as they may be at increased risk of developing adverse events. Veterans with renal disease/impairment, hepatic disease/impairment, cardiac illness (e.g. coronary vascular disease, congestive heart failure), or hypokalemia at screening will also be excluded. Since mifepristone use can prolong the corrected QT (QTc) interval in a dose-related manner, Veterans with a prolonged QTc interval, defined as >450 msec, on the ECG at screening will be excluded. To evaluate QTc prolongation post-mifepristone treatment, an ECG will also be performed at both the 3 day follow up visit (visit 1.5) and 1 week follow-up visit (week 1, visit 2).

Participants on potent CYP3A4 inhibitors (fluconazole, ketoconazole, itraconazole, erythromycin, rifampin) and some anticonvulsants (e.g., phenytoin, phenobarbital, and carbamazepine) will be excluded since these medications impact the metabolism of mifepristone (see Risk/Benefit Assessment for details). Due to an increased risk of adverse drug reactions, Veterans taking simvastatin, lovastatin, fentanyl, pimozide, bupropion, nefazodone, dihydroergotamine, ergotamine, quinidine, sirolimus, carvedilol, propanolol, diltiazem, verapamil or tacrolimus will also be excluded. Since the impact of mifepristone on the male reproductive system has not been extensively studied, only Veterans willing to use effective means of birth control for up to 90 days after mifepristone ingestion will be eligible; this will cover the critical period of fetal development.

Psychotropic medication use is exclusionary at study entry; Veterans who have been previously treated with a stable regimen may not be enrolled until a minimum of five half-lives have elapsed since the Veteran last took any psychotropic medications. (Sleep aids such as trazodone (up to 50 mg/day) or zolpidem (up to 10 mg/day) may be offered to Veterans with insomnia on an as-needed basis at the onset of the study.) Major depression and other anxiety disorders are not exclusionary since they frequently co-occur with PTSD and it remains unclear whether their presence represents true comorbidity, symptom overlap, or severe illness. Since mild head trauma is common in the military population in general, excluding such participants would diminish the generalizability of the sample; participants with severe traumatic brain injury (TBI), defined as an extended period of unconsciousness or amnesia following injury, will be excluded. The Ohio State University (OSU) TBI Identification Method will be used to assess lifetime history of TBI. This method first establishes all significant injuries in one's life and then determines if a TBI may have occurred based on whether the participant experienced a loss of consciousness (LOC) and, if so, for how long. A person is said to have a mild TBI if LOC does not exceed 30 minutes for any injury, a moderate TBI if LOC is between 30 minutes and 24 hours, and a severe TBI if LOC exceeds 24 hours. The OSU TBI assessment will be administered by a trained rater during the psychiatric evaluation conducted at screening.

Additionally, Veterans diagnosed with alcohol/substance abuse and dependence will be excluded only if they are recently engaged in a maladaptive pattern of use or abuse. More specifically, persons who meet diagnostic criteria for alcohol/substance dependence will be excluded if they have manifested dependence within the previous three months (i.e., have met three or more of the seven criteria for a maladaptive pattern of use in the last three months). Persons with alcohol/substance abuse (who, by definition, do not meet criteria for alcohol dependence) will be excluded if they have shown a maladaptive pattern of alcohol use during the past one month (i.e., have met one or more of the four criteria for a maladaptive pattern of abuse).

Veterans who are currently receiving psychotherapies - individually or in a group setting - that are considered to have significant benefit for PTSD, according to the VA and Department of Defense (DoD's) Treatment Guidelines, will also be excluded. These therapies are cognitive therapy for PTSD (e.g. cognitive processing therapy (CPT)), exposure therapy (e.g., prolonged exposure therapy), stress inoculation training, and eye movement desensitization and reprocessing (EMDR). Other forms of therapy and case management which do not specifically target PTSD symptoms and/or have not been shown to provide significant benefit in PTSD will be allowed at entry and throughout the study (e.g. supportive therapy, psychodynamic therapy, anger management, cognitive behavioral therapy for symptoms or problems other than PTSD).

The investigators recognize that PTSD in women is increasingly common and effective treatments are needed for this group as well. However, women will be excluded from this initial trial for safety reasons, since mifepristone is an abortifacient. Should mifepristone prove to be effective in male Veterans with PTSD, this would provide a rationale for future studies in women, employing additional safeguards.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male veteran.
* Veteran meets the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnostic criteria for chronic PTSD.
* Veteran has a CAPS total score (past month symptom status) greater than or equal to 50 at screening.
* For veterans taking psychotropic medications (i.e., antidepressants, antipsychotics or anxiolytics/sedative-hypnotics), the veteran will be on a stable dose for at least five weeks prior to screening.
* For veterans not taking psychotropic medication, a minimum of five half-lives must elapse prior to screening since the veteran last took any given psychotropic medication.

Exclusion Criteria:

* Veteran recently continued to engage in a maladaptive pattern of alcohol/substance use and/or abuse (as defined in protocol).
* Veteran has used potent CYP3A4 inhibitors (fluconazole, ketoconazole, itraconazole, erythromycin, rifampin) and inducers within five half-lives prior to randomization.
* Veteran is taking simvastatin, lovastatin, fentanyl, pimozide, bupropion, nefazodone, dihydroergotamine, ergotamine, quinidine, sirolimus, tacrolimus, or clarithromycin, cyclosporine, St. John's Wort, diltiazem, verapamil, propranolol, alprazolam, carvedilol or some anticonvulsants (phenytoin, phenobarbital, or carbamazepine) within five half-lives prior to randomization.
* Veteran is taking oral corticosteroids within five half-lives prior to randomization.
* Veteran should be free of a major medical illness and medical condition that contraindicate the administration of mifepristone. These include but are not limited to:

  1. Veteran has a history of adrenal insufficiency or a low plasma cortisol level at screening (a.m. level less than 5 mcg/dl or a p.m. level of less than 3 mcg/dl.)
  2. Veteran has a history of severe traumatic brain injury, a history of a stroke, or another neurological illness or injury likely to impact cognitive functioning.
  3. Veteran has diabetes mellitus, an endocrinopathy, or another major medical illness.
  4. Veteran has a history of cardiovascular disease including a history of angina, myocardial infarction or other evidence of coronary artery disease, or congestive heart failure.
  5. Veteran has prolonged QTc interval >450 msec on ECG at screening.
  6. Veteran has hypokalemia at screening (defined as potassium level < 3.5 Milliequivalent Per Liter (mEq/L)).
  7. Veteran has a history of hepato-biliary disease or an aspartate transaminase (AST), alanine transaminase (ALT) greater than 2 times the Upper Limit of Normal (ULN).
  8. Veteran has a history of renal disease or an estimated glomerular filtration rate (GFR) of < 60 ml/min.
* Veteran has a lifetime diagnosis of schizophrenia, schizoaffective disorder, or type I bipolar disorder.
* Veteran has a history of attempted suicide within the previous two years or active suicidal ideation within the past month as assessed by the Columbia-Suicide Severity Rating Scare (C-SSRS).
* Veteran is currently receiving specialized trauma-focused psychotherapy, such as prolonged exposure therapy and cognitive processing therapy.
* Veteran is not willing to use effective means of birth control during the study.
* Veteran has a history of allergic reaction to mifepristone.
* Veteran is found to be unsuitable for study participation at the discretion of the site investigator for any reason.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Golier, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (5):
- United States (5):
  - VA San Diego Healthcare System, San Diego, California
  - Albuquerque VA Medical Center, Albuquerque, New Mexico
  - James J. Peters VA Medical Center, The Bronx, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Golier JA, Li X, Bizien M, Hurley RA, Bechard BW, Kimbrell T, Flory JD, Baker DG, Yehuda R, Reda DJ. Efficacy and Safety of Mifepristone in the Treatment of Male US Veterans With Posttraumatic Stress Disorder: A Phase 2a Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2310223. doi: 10.1001/jamanetworkopen.2023.10223. PMID 37159200

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone (600 mg/Day): 600 mg/day mifepristone for one week
  Mifepristone (600 mg/day) or placebo (sugar pill): 600 mg/day mifepristone or placebo (sugar pill) for one week
- Sugar Pill: Placebo (sugar pill) for one week
  Mifepristone (600 mg/day) or placebo (sugar pill): 600 mg/day mifepristone or placebo (sugar pill) for one week
Period: Overall Study
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Started | 41 | 40
Completed | 34 | 35
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 7 | 4
Not completed — Ineligible patient randomized | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline comparison is based on 80 randomized patients who satisfied all study entry criteria and received at least one dose of study medication. The one subject (placebo group) who was found to be ineligible after randomization and was terminated in study dosing phase was not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [33 to 53] | 37 [30 to 56] | 40 [31 to 55.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 39 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 11 | 25
  White | 20 | 26 | 46
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Clinical Responders at 4-week Follow-up
Description: A clinical responder at 4-week is defined as a participant who achieves a 30% or greater reduction in CAPS total score (past week symptom status) from baseline to 4-week follow-up. The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. The CAPS total score (ranges 0 - 136) is the sum of 17 PTSD symptoms (each symptom is the sum of the frequency score (ranges 0-4) and the intensity score (ranges 0-4)) in the three different symptom subcategories (intrusive/re-experiencing (0-40), avoidance/numbing (0-56) and hyperarousal (0-40)). The higher is the CAPS total score, the worse is the PTSD symptom. Higher percentage of responders indicate a better drug effect in treating PTSD symptoms.
Time Frame: week 4
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 4-week CAPS assessment were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 39 | 38
Participants
  ≥ 30% Reduction in CAPS Total Score | 15 | 12
  < 30% Reduction in CAPS Total Score | 24 | 26

2. Secondary Outcome: Percentage of Clinical Responders at 12-week Follow-up (End of Study)
Description: A clinical responder at 12-week is defined as a participant who achieves a 30% or greater reduction in CAPS total score (past week symptom status) from baseline to 12-week follow-up. The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. The CAPS total score (ranges 0 - 136) is the sum of 17 PTSD symptoms (each symptom is the sum of the frequency score (ranges 0-4) and the intensity score (ranges 0-4)) in the three different symptom subcategories (intrusive/re-experiencing (0-40), avoidance/numbing (0-56) and hyperarousal (0-40)). The higher is the CAPS total score, the worse is the PTSD symptom. Higher percentage of responders indicate a better drug effect in treating PTSD symptoms.
Time Frame: week 12
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 12-week CAPS assessment were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 32 | 35
Participants
  ≥ 30% Reduction in CAPS Total Score | 10 | 14
  < 30% Reduction in CAPS Total Score | 22 | 21

3. Secondary Outcome: Change in CAPS Total Score From Baseline to 4-week and 12-week
Description: The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. The CAPS total score ranges 0 to 136, which is the sum of 17 PTSD symptoms (each symptom is the sum of the frequency score (ranges 0-4) and the intensity score (ranges 0-4)) in the three different symptom subcategories (intrusive/re-experiencing (0-40), avoidance/numbing (0-56) and hyperarousal (0-40)). A higher CAPS total score indicates worse PTSD symptoms. A positive change score indicates an increased CAPS total score (i.e., worse PTSD symptoms) at 4-week (12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-week
Population: Participants in the modified intent-to-treat (mITT) population were analyzed. This includes 80 randomized participants who took at least a single dose of study medication and met all study eligibility criteria. Mean and 95% Confidence Interval (CI) reported is the least square estimates from the repeated-measures analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -13.96 [-19.61 to -8.31] | -15.83 [-21.57 to -10.08]
  Change Score from Baseline to 12-week | -15.15 [-22.34 to -7.96] | -18.06 [-25.16 to -10.96]

4. Other Pre Specified Outcome: Change in CAPS Intrusive Symptom Scores From Baseline to 4-Week and 12-Week
Description: The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. Its intrusive symptom subscale (ranges 0 - 40) is the sum of 5 PTSD symptoms (each ranges 0 - 8) in the intrusive/re-experiencing symptom subcategory. A higher intrusive symptom score indicates worse PTSD symptoms. A positive change score indicates an increased intrusive symptom score (i.e., worse PTSD symptoms) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-Week and 12-Week
Population: Participants in the modified intent-to-treat (mITT) population were analyzed. This includes 80 randomized participants who took at least a single dose of study medication and met all study eligibility criteria. Mean and 95% CI reported is the least square estimates from the repeated-measures analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mifepristone (600 mg/Day): 600 mg/day mifepristone for one week Mifepristone (600 mg/day) or placebo (sugar pill): 600 mg/day mifepristone or placebo
- Sugar Pill: Placebo (sugar pill) for one week
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -4.27 [-6.89 to -1.64] | -5.49 [-8.17 to -2.82]
  Change Score from Baseline to 12-week | -4.77 [-7.91 to -1.63] | -7.78 [-10.86 to -4.70]

5. Other Pre Specified Outcome: Change in CAPS Avoidance Symptom Scores From Baseline to 4-Week and 12-Week
Description: The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. Its avoidance symptom subscale (ranges 0 - 56) is the sum of 7 PTSD symptoms (each ranges 0 - 8) in the avoidance/emotional numbing symptom subcategory. A higher avoidance symptom score indicates worse PTSD symptoms. A positive change score indicates an increased avoidance symptom score (i.e., worse PTSD symptoms) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
  The higher is the avoidance/emotional numbing PTSD subscale score, the worse is the PTSD symptom.
Time Frame: baseline to 4-Week and 12-Week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mifepristone 600 mg/Day: 600 mg/day mifepristone for one week
Arm/Group | Mifepristone 600 mg/Day | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -6.24 [-9.24 to -3.24] | -6.81 [-9.86 to -3.76]
  Change Score from Baseline to 12-week | -6.30 [-9.99 to -2.60] | -6.22 [-9.87 to -2.57]

6. Other Pre Specified Outcome: Change in CAPS Hyperarousal Symptom Scores From Baseline to 4-Week and 12-Week
Description: The Clinical Administered PTSD Scale (CAPS) was used to assess the diagnosis of PTSD symptoms. Its hyperarousal symptom subscale (ranges 0 - 40) is the sum of 5 PTSD symptoms (each ranges 0 - 8) in the hyperarousal symptom subcategory. A higher hyperarousal symptom score indicates worse PTSD symptoms. A positive change score indicates an increased hyperarousal symptom score (i.e., worse PTSD symptoms) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-Week and 12-Week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mifepristone (600 mg/Day): 600 mg/day mifepristone for one week
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -3.35 [-5.16 to -1.53] | -3.49 [-5.33 to -1.64]
  Change Score from Baseline to 12-week | -3.22 [-5.37 to -1.08] | -4.15 [-6.24 to -2.05]

7. Other Pre Specified Outcome: Change in Depression (Measured by the BDI Total Score) From Baseline to 4-Week and 12-Week
Description: The Beck Depression Inventory (BDI) total score (ranges 0-63) is the sum of 21 items (each item rated on a 4-point scale of 0 to 3) relating to symptoms of depression, cognitions, and physical symptoms. The BDI total score measures the overall severity of depression. The higher the BDI total score, the more severe the depression. A positive change score indicates an increased BDI total score (i.e., more severe depression) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-Week and 12-Week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -3.50 [-6.20 to -0.79] | -4.52 [-7.29 to -1.75]
  Change Score from Baseline to 12-week | -2.25 [-5.34 to 0.83] | -5.07 [-8.19 to -1.96]

8. Other Pre Specified Outcome: Changes in PTSD Symptom Severity (Measured by the Stressful Life Total Score From the PTSD Checklist) From Baseline to 4-Week and 12-Week
Description: Stressful life total score (ranges 17-85) is the sum of the severity ratings of the 17 PTSD-related symptoms (each symptom is rated on a 5-point scale of 1=not at all to 5=extremely) over the past week. It evaluates the extent to which responders have been "bothered" by the symptoms of PTSD. The higher stressful life score indicates more stressful life events. A positive change score indicates an increased stressful life total score (i.e., more stressful life events) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-Week and 12-Week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -6.84 [-9.90 to -3.78] | -8.65 [-11.80 to -5.49]
  Change Score from Baseline to 12-week | -6.84 [-10.54 to -3.14] | -8.12 [-11.90 to -4.34]

9. Other Pre Specified Outcome: Change in Sleep Quality (Measured by the PSQI Total Score) From Baseline to 4-Week and 12-Week
Description: The Pittsburgh Sleep Quality Index (PSQI) assesses self-report sleep quality and disturbances. Nineteen individual items generate 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. Each component is scored from 0=better to 3=worse. The sum of the 7 component scores yields the PSQI total score (range 0-21) with a higher score indicating a worse sleep quality. A positive change score indicates an increased PSQI total score (i.e., worse sleep quality) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: baseline to 4-Week and 12-Week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -1.63 [-2.67 to -0.59] | -1.27 [-2.34 to -0.21]
  Change Score from Baseline to 12-week | -0.86 [-2.10 to 0.40] | -2.04 [-3.29 to -0.79]

10. Other Pre Specified Outcome: Change in Anger Level (Measured by the STAXI Total Score) From Baseline to 4-Week and 12-Week
Description: The State-Trait Anger Expression Inventory (STAXI) total score is the sum of 10 items assessing intensity of anger as an emotional state (State Anger) and the disposition to experience angry feelings as a personality trait (Trait Anger). Each item consists of a 4-point scale (1=not at all, 4=very much) that assess intensity of anger at a particular moment and the frequency of anger experience, expression and control. The STAXI total score ranges from 10 to 40, with a higher score indicating a higher intensity of anger.The sum of the 7 component scores yields the PSQI total score (range 0-21) with a higher score indicating a worse sleep quality. A positive change score indicates an increased STAXI total score (i.e., higher intensity of anger) at 4-week (or 12-week) compared to its baseline value, while a negative change score indicates an opposite direction.
Time Frame: Baseline to 4-week and 12-week
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 39
units on a scale
  Change Score from Baseline to 4-week | -0.61 [-2.78 to 1.56] | -1.83 [-4.05 to 0.40]
  Change Score from Baseline to 12-week | -1.73 [-3.85 to 0.39] | -3.20 [-5.32 to -1.08]

11. Other Pre Specified Outcome: Change in Plasma Cortisol From Baseline to 1-Week
Description: Mifepristone will induce acute increase in Cortisol and ACTH levels. Higher Cortisol value indicates higher magnitude of mifepristone's effects on negative feedback inhibition. Cortisol value in placebo group at follow-up visits will remain at the similar level as its baseline magnitude. A positive change value indicates increased cortisol level at 1-week (i.e., higher magnitude on negative feedback inhibition) compared to its baseline value, while a negative change value indicates an opposite direction.
Time Frame: Baseline to 1-week
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 1-week blood collection on cortisol were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Median (Inter-Quartile Range); unit: ug/dl
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 38
ug/dl | 22.3 [3.3 to 33.2] | -0.9 [-3.4 to 3.6]

12. Other Pre Specified Outcome: Change in Plasma Cortisol From Baseline to 4-Week
Description: Mifepristone will induce acute increase in Cortisol and ACTH levels. Higher Cortisol value indicates higher magnitude of mifepristone's effects on negative feedback inhibition. Cortisol value in placebo group at follow-up visits will remain at the similar level as its baseline magnitude. A positive change value indicates an increased cortisol level at 4-week (i.e., higher magnitude on negative feedback inhibition) compared to its baseline value, while a negative change value indicates an opposite direction.
Time Frame: Baseline to 4-week
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 4-week blood collection on cortisol were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Median (Inter-Quartile Range); unit: ug/dl
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 38 | 35
ug/dl | -0.6 [-7.0 to 3.1] | -0.4 [-2.4 to 3.4]

13. Other Pre Specified Outcome: Change in Adrenocorticotropic Hormone (ACTH) From Baseline to 1-week
Description: Mifepristone will induce acute increase in Cortisol and ACTH levels. Higher ACTH value indicates higher magnitude of mifepristone's effects on negative feedback inhibition. ACTH value in placebo group at follow-up visits will remain at the similar level as its baseline magnitude. A positive change value indicates an increased ACTH level at 1-week (i.e., higher magnitude on negative feedback inhibition) compared to its baseline value, while a negative change value indicates an opposite direction.
Time Frame: baseline to 1-week
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 1-week blood collection on ACTH were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 41 | 38
pg/ml | 28.8 [7.9 to 63.7] | -0.5 [-5.0 to 5.4]

14. Other Pre Specified Outcome: Change in Adrenocorticotropic Hormone (ACTH) From Baseline to 4-week
Description: Mifepristone will induce acute increase in Cortisol and ACTH levels. Higher ACTH value indicates higher magnitude of mifepristone's effects on negative feedback inhibition. ACTH value in placebo group at follow-up visits will remain at the similar level as its baseline magnitude. A positive change value indicates an increased ACTH level at 4-week (i.e., higher magnitude on negative feedback inhibition) compared to its baseline value, while a negative change value indicates an opposite direction.
Time Frame: Baseline to 4-week
Population: Participants who were included in the modified intent-to-treat (mITT) population and also did not miss 4-week blood collection on ACTH were analyzed. The mITT population include participants who took at least a single dose of study medication and also met all study eligibility criteria.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
Number analyzed (Participants) | 38 | 35
pg/ml | -0.8 [-7.3 to 2.6] | 1.5 [-5.5 to 6.2]

ADVERSE EVENTS:
Time Frame: Participants were enrolled for 3 months. Adverse Events (AE) and Serious Adverse Events (SAE) information were collected from randomization to study medication/placebo until 12 week follow-up and/or participant termination (whichever occurred first). If a participant experienced more than 1 of a given AE, the participant was counted only once for that AE. If a participant experienced more than one AE in a system organ class (SOC), the participant was counted only once in that SOC.
Arm/Group | Mifepristone (600 mg/Day) | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/40
Other Adverse Events (participants affected / at risk) | 21/41 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (600 mg/Day) (N=41) | Sugar Pill (N=40)
Social stay hospitalization (Social circumstances) | 1 (1) | 0 (0) — This participant developed homicidal ideation in the setting of family stress and homelessness, which resulted in psychiatric hospitalization (preferred term: Social stay hospitalization). This event was not related to the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (600 mg/Day) (N=41) | Sugar Pill (N=40)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) — not related to study drug
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Energy Increased (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) — not related to study drug
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — not related to study drug
Blood thyroid stimulating hormone increase (Investigations) | 1 (1) | 0 (0)
Electrocardiogram Prolonged QT interval (Investigations) | 1 (2) | 2 (2)
Glomerular Filtration Rate Decrease (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0) — not related to study drug
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) — not related to study drug
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — not related to study drug
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Exertional headache (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 1 (1)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — not related to study drug
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) — 1 rash (mifepristone) and 1 rash (placebo) were not related to study drug
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sympathectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — not related to study drug
Hypertension (Vascular disorders) | 2 (2) | 0 (0) — 1 hypertension (mifepristone) was not related to study drug
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study only look at a low dose of mifepristone (600 mg /day) for a short period (7 days). A higher dose of mifepristone (900 mg, 1200mg and etc.) haven't been studied in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes